CLINICAL TRIAL: NCT03158350
Title: A Tooth Brushing Technique That Reduces Gingival Inflammation and Toothbrush Deformation
Brief Title: Toothbrush Wear and Its Effect on Subgingival Inflammation Using Two Different Brushing Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11724
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Gingival Inflammation
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stationary Bristle Technique (SBT) (Experimental): Instructed brushing method. Participants are asked to brush twice daily, for 2 minutes at a time, following instructions for the Stationary Bristle Technique.
  Interventions: Other: Instructed Brushing Method
- Non-Stationary Bristle Technique (NSBT) (No Intervention): The control group will be asked to brush twice daily, for 2 minutes at a time, following their normal toothbrushing technique.

INTERVENTIONS:
Other: Instructed Brushing Method — Stationary Bristle Technique
  Arms: Stationary Bristle Technique (SBT)

SUMMARY:
Toothbrush plaque removal, along with interproximal flossing, helps to maintain the oral cavity free from periodontal diseases and dental caries. Although techniques such as the Bass Technique (BT), the Modified Bass Technique (MBT) and the Modified Stillman Technique (MST) are taught to dental students, dental hygiene students, and dental assistants, there is little evidence to discern which technique is more effective in reducing or preventing gingival inflammation.

At Tufts University School of Dental Medicine (TUSDM), a modification of the Bass intrasulcular technique is advocated to many students. We call this modification of the Bass technique a Stationary Bristle Technique (SBT), which is an intrasulcular technique that maintains the toothbrush bristle ends essentially stationary on the tooth cervically and in the gingival crevice.

In this study, half of the participants were taught the Stationary Bristle Technique Group, while the other half were not be provided with instructions, but asked to brush as normal (non-interventional group) throughout the duration of the study.

DETAILED DESCRIPTION:
This is a double-armed, randomized clinical trial. The primary aim of this study is to compare whether a Stationary Brushing Technique (SBT) is more effective in the reduction of gingival inflammation than permitting people to brush the way they normally do without instruction (Non-Stationary Brushing Technique).

Gingival inflammation is evidenced by the percentage (%) sites with Bleeding on Probing (BoP). The primary time-point will be at 4 weeks.

The amount of toothbrush bristle deformation at 4 weeks, 12, and 16 weeks of brushing with a SBT and with a NSBT will also be evaluated. 3. The secondary evaluation of BoP will be at the 12 and 16 week time-point.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Subjects must have at least 20 teeth
* Subjects must have had a professional dental prophylaxis done in the 3 months prior to the beginning of the study
* Subjects exhibiting 10% or greater BoP at the baseline examination

Exclusion Criteria:

* Subjects wearing fixed orthodontic appliances (including lingual retainers or Invisalign®)
* Subjects who smoke (=more than 0 cigarettes a day)
* Subjects who received antibiotic treatment during the month prior to the beginning of the study
* Subjects who have cervical probing depth (PD) greater than 3mm
* Subjects diagnosed with periodontal disease at any site as defined bleeding on probing with cervical probing depths greater than 3 mm and loss of cervical attachment.
* Subjects who are currently pregnant (self-report).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Gingival Inflammation | From Baseline up to 4 weeks
  Measured by the percentage of sites with BoP. The percentage of sites with BoP at each time point will be calculated by group

SECONDARY OUTCOMES:
Toothbrush Bristle Deformation | From baseling up to 16 weeks
  Toothbrush bristle deformation will be measured at 4 weeks, 12 weeks, and 16 weeks of brushing with SBT or NSBT. The mean and standard deviation of the deformation measurements (length and width) will be calculated at each time point for each group.
Change in BoP | From baseline up to 16 weeks
  The secondary evaluation of BoP will be at the 12 and 16 week time-point.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Levi, Jr., DMD, Principal Investigator — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No